CLINICAL TRIAL: NCT05069818
Title: Variance of HRD From Primary to Recurrent in High-grade Serous Ovarian Cancer
Brief Title: Variance of HRD From Paired Ovarian Cancer
Acronym: HOPEII
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiaoxiang Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaoxiang Chen, Academic secretary of gynecological oncology Committee of Jiangsu anti cancer association, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Other Study IDs: JiangsuCIH011
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Ovarian Cancer; HRD; Platinum-sensitive Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The formalin fixation and paraffin embedding (FFPE ) samples from the primary and secondary cytoreductive surgery will be obtained after patients' informed consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Homologous recombination deficiency (HRD) is an important biomarker of poly (ADP-ribose) polymerase inhibitor (PARPi) in patients with high-grade serous ovarian cancer (HGSOC). The stability of HRD in the recurrent HGSOC and its primary pair remains unknown.

DETAILED DESCRIPTION:
This study intends to perform HRD testing of ovarian cancer in the recurrent HGSOC and its primary pair, furtherly correlate HRD status and clinical characteristics in the recurited population.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects join the study voluntarily and sign informed consent;
2. Female subjects are older than 18 years;
3. ECOG(Eastern Cooperative Oncology Group) physical status score is 0-2;
4. Life expectancy≥3 months;
5. Histologically confirmed FIGO(International Federation of Gynecology and Obstetrics ) III/IV ovarian cancer, fallopian tube cancer, or primary peritoneal cancer; Participants must have high-grade serous histology

Exclusion Criteria:

1. Personnel involved in the formulation or implementation of the research plan;
2. The subjects had other malignant diseases in past 2 years, except skin squamous cell carcinoma, basal-like carcinoma, breast intraductal carcinoma in situ, or cervical carcinoma in situ;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Platinum-sensitive relapsed high-grade serous ovarian cancer patients undergoing secondary cytoreductive surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Loss of heterozygosity (LOH) score in the primary and recurrent ovarian cancer | Through study completion, an average of 1 year]
  The LOH score is a scale describing the genomic loss of heterozygosity status in the primary or recurrent tumor of an ovarian cancer patient. The score is determined by analyzing more than 3500 SNPs spaced at 1Mb intervals across the genome on the FoundationOne CDx test and extrapolating an LOH profile, excluding arm and chromosome-wide LOH segments. The score is summarized as the percentage of the genome with LOH regions.
Homologous recombination deficiency (HRD) status | Through study completion, an average of 1 year
  The HRD status for primary or recurrent tumor in a patient is considered according to the LOH score and genomic mutation status of BRCA1 and BRCA2 genes in the sample. A sample with LOH≥16%，and/or with genomic mutation in BRCA1 or BRCA2 gene, is defined as HRD positive. Otherwise, a sample with LOH<16% and wild type BRCA1/BRCA2 genes is defined as HRD negative.

SECONDARY OUTCOMES:
Progression-free survival | From the beginning of the patient's onset, an average of 1 year
  Progression-free survival in recruited patients
Overall survival | From the beginning of the patient's onset, an average of 3 year
  Overall survival in recruited patients

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxiang Chen Chen, MD,PhD, Study Chair — Jiangsu Cancer Institute & Hospital
Locations (1):
- Xiaoxiang Chen, Nanjing, Jiangsu, China